CLINICAL TRIAL: NCT06374719
Title: WiTNNess: An International Natural History Study of Autosomal Recessive TNNT1 Myopathy
Brief Title: WiTNNess - TNNT1 Myopathy Natural History Study
Acronym: WiTNNess
Status: Recruiting | Type: Observational
Sponsor: Clinic for Special Children (Other)
Responsible Party: Sponsor
Other Study IDs: WiTNNess
Record Dates: First submitted 2024-04-12; First posted 2024-04-19 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: TNNT1-associated Myopathy; Infantile-onset Nemaline Rod Myopathy; Myopathies, Nemaline; Myopathy; Myopathy, Rod; Myopathy; Hereditary; Amish Nemaline Myopathy; Nemaline Myopathy 5; NEM5; Genetic Muscle Disease; Recessive Hereditary Disorder (Autosomal); ANM
MeSH Terms: conditions — Myopathies, Nemaline; Muscular Diseases; Nemaline myopathy 5

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective: Participants in the prospective cohort are enrolled during early infancy, shortly after diagnosis, and followed longitudinally with repeated assessments until reaching the primary study outcome.
- Cross-Sectional: Participants in the cross-sectional cohort enroll at any time after diagnosis and all study data are collected at a single time point.

SUMMARY:
WiTNNess is designed to accurately document the natural course and variation of muscle disease caused by pathogenic changes of the TNNT1 gene. The primary aim of the study is to specify meaningful outcome measures for future clinical trials. WiTNNess is open to children and adults worldwide. Participants can choose to include their information once (cross-sectional cohort) or every few months (prospective cohort).

DETAILED DESCRIPTION:
WiTNNess is an observational study that includes prospective and cross-sectional arms, both of which include people diagnosed with autosomal recessive TNNT1-associated muscle disease, commonly described as a form of infantile-onset (NEM5A) or childhood-onset (NEM5B) nemaline rod myopathy. The study's primary objective is to establish the nature and time course of disease outcomes under current treatment, so that these can later be compared to outcomes achieved with novel disease-modifying therapies (i.e., interventional trials).

Participants from all over the world are welcome to enroll in either arm of the WiTNNess study. Following appropriate consent, those in the prospective arm are followed long-term. Recurring assessments are performed at the participant's home, the Clinic for Special Children, or a partnering clinical site, depending on the individual's particular circumstances. Basic assessments include vital signs, a physical exam, documentation of motor milestones, growth measurements, and blood chemistry values. Participant's may also undergo non-invasive ultrasound of the heart (echocardiogram) and one or more chest radiographs.

Participants in the cross-sectional arm are contacted once after consent. Members of the WiTNNess study team partner with healthcare providers and family members to capture pertinent medical history, physical exam findings, growth metrics, and motor milestones at the time of contact.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with biallelic pathogenic variants of TNNT1
* Infantile-onset or childhood-onset proximal weakness without confounding medical conditions that could effect muscle health.

Exclusion Criteria:

* Another known or suspected medical condition (genetic or acquired) that could potentially alter the natural disease course or otherwise interfere with completion of study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes anyone diagnosed with biallelic pathogenic variants of TNNT1
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-09-23 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | Day 1 up to 15 years
  The primary outcome is time until death or permanent ventilatory support, defined as any invasive (e.g., tracheostomy) or non-invasive (e.g., bilevel positive airway pressure) mechanical ventilatory assistance for ≥16 hours daily during ≥14 consecutive days in the absence of a reversible clinical state.

SECONDARY OUTCOMES:
Motor Milestones | All milestones normally achieved by postnatal age 17.1 months (normal 99th percentile reference value for independent walking).
  Six motor milestones that include sitting without support, standing with assistance, hands and knees crawling, walking with assistance, standing alone, and walking alone, as defined by the Word Health Organization Multicentre Growth Reference Study.
Thriving | Day 1 up to 15 years
  Maintain weight at ≥3rd WHO reference percentile for sex and age. The ability to swallow normally and maintain body weight equal to or greater than the WHO 3rd reference percentile for sex and age without requiring non-oral feeding support (i.e., nasogastric or gastrostomy tube).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Strauss, MD, Principal Investigator — Clinic for Special Children
Locations (1):
- Clinic for Special Children, Gordonville, Pennsylvania, United States